CLINICAL TRIAL: NCT03625973
Title: Creating Physical Objects With 3D Printers to Stimulate Reminiscing for Memory Loss [2 R44 AG049548-02A1]
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Moai Technologies LLC (Other)
Collaborators: St. Louis University (Other); The University of Texas at Arlington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MoaiTech
Record Dates: First submitted 2018-07-16; First posted 2018-08-10 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Dementia
Keywords: Dementia; Memory, Episodic; Printing, Three-Dimensional
MeSH Terms: conditions — Dementia; Recurrence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A social work graduate assistant from Dr. Berg-Weger's program and Dr. Anderson's program will administer the various behavioral tests that will produce the outcome measures. This will be a different individual than the graduate assistants who conduct the RT sessions with participants. Also the assistant administering the tests will be blind as to the treatment assignment of the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 16 Weeks of 3D-RT (Experimental): Participants will receive 16 weeks of Reminiscence Therapy using 3D printed objects as stimuli.
  Interventions: Behavioral: 3D-RT
- 8 Weeks of 3D-RT (Experimental): Participants will receive 8weeks of Reminiscence Therapy using 3D printed objects as stimuli and 8 weeks of RT using verbal stimuli.
  Interventions: Behavioral: 3D-RT
- 16 Weeks of RT using Verbal Stimuli (Active Comparator): Participants will receive 16 weeks of RT using verbal stimuli to reminiscence.
  Interventions: Behavioral: RT-Verbal

INTERVENTIONS:
Behavioral: 3D-RT — Objects printed using 3D printing media will be used as stimuli in Reminiscence Therapy
  Arms: 16 Weeks of 3D-RT; 8 Weeks of 3D-RT
Behavioral: RT-Verbal — Verbal cues will be used as stimuli in Reminiscence Therapy
  Arms: 16 Weeks of RT using Verbal Stimuli

SUMMARY:
In 2013 an estimated 5 million people age 65 and older had Alzheimer's disease. Longer life spans and aging baby boomers will cause this number to grow rapidly. More than 50% of residents in assisted living and nursing homes have some form of dementia or cognitive impairment and the number is increasing every day.

As a form of person-centered, non-pharmacological dementia care, Reminiscence Therapy (RT) holds considerable promise. Improvements in mood, quality of life, social interaction, cognition, memory and a reduction in caregiver stress have been noted. This project will develop an operational model for identifying and producing 3D personal objects using 3D printing technology, and deploying them for use in RT. The research also will evaluate the effectiveness of using 3D-printed objects in RT compared to other types of memory stimuli. This novel approach to the "personalization" of reminiscence therapy will result in better social and mental health outcomes for individuals with dementia.

DETAILED DESCRIPTION:
Objective:

The objective of the field evaluation is to determine the effectiveness of reminiscence therapy (RT) using replicas of personal objects produced by 3D printing. To address this objective, randomized control field trials will be conducted in which the effects of high and low doses of RT using 3D-printed objects will be compared to the effects of using only traditional verbally-presented stimuli during RT. Effects will be measured on autobiographical memory, psycho-social status, and quality of life.

Participants:

The Co- Investigators, Dr. Berg-Weger and Dr. Anderson, in cooperation with the participating care organizations, will identify a total of 156 persons with memory loss of varying gender, race, and ethnicity to participate in the field trial.

Study Design and Implementation:

Two hypotheses will be tested. Hypothesis 1. An RT program dose consisting of 16 weeks of RT sessions using personalized physical objects produced by 3D printing will result in more and richer autobiographical reminiscence than a 16 week RT program dose consisting of 8 weeks of RT sessions using personalized 3D objects followed by 8 weeks of RT using verbal stimuli. Further, it is hypothesized that a full 16 weeks of RT using 3D objects will have a more significant positive effect on overall cognitive functioning, communication, and quality of life than 8 weeks of RT using 3D objects plus 8 weeks of RT using verbal memory stimuli.

Hypothesis 2. Both programs of RT using personalized physical 3D-printed objects will result in significantly greater and richer autobiographical reminiscence than a program consisting of 16 weeks of more traditional RT using verbal memory stimuli, and also have a positive effect on overall cognitive functioning, communication, and quality of life.

Study Design:

A between groups design will be used to examine these hypotheses, with participants assigned randomly to one of three groups:

1. a High Dose group receiving RT using personalized 3D objects for 16 weeks,
2. a Low Dose group receiving RT using personalized 3D objects for 8 weeks followed by 8 weeks of RT using traditional verbal stimuli, or
3. a control group receiving more traditional RT using verbal stimuli related to personal objects of interest.

The proposed high and low RT dosages are based on the higher and lower range dosages reported in two recent meta-analyses of RT. Personalized 3D objects will be identified for 3D-RT group participants by the therapist using a mobile application developed specifically for this project. Verbal stimuli for RT for the traditional RT group will be developed using exactly the same life history questions used in the mobile application. Questions will be selected from the list and discussed, one by one, until the discussion leads to a topic being identified by the Person With Memory Loss (PWML). An effort will be made to ensure that this process of identifying verbal stimuli for the Verbal RT group participants involves therapist contact time equivalent to that expended by the therapist in identifying personalized 3D objects for 3D-RT group participants.

Thirty-minute therapy sessions will be conducted 1 time each week for 16 weeks. Every two weeks, a new 3D object will be identified by the caregiver/therapist working with the PWML, printed by Moai Technologies, and introduced to the therapy. Thus, each object or topic will serve as the RT stimulus for two sessions. In the unlikely event that the 3D object does not stimulate a full 30 minutes of discussion, the therapist will be prepared with more general reminiscence topics to introduce so that a full 30-minute session can be completed and contact time across sessions held constant. Participating RT therapists will be trained on how to make the transition. For those in the Verbal-RT group, a new verbally-presented topic of autobiographical interest to the PWML will be identified and introduced every two weeks. As with the 3D object groups, if the identified topic does not stimulate a full 30 minutes of discussion, the therapist will be prepared with more general reminiscence topics to introduce so that a full 30-minute session can be completed.

This approach to delivering RT by means of regular, structured sessions with a trained caregiver draws on the successful paradigm developed in the United Kingdom for Individual Cognitive Stimulation Therapy (CST). Notably, all project collaborators in the St. Louis area are part of the university's CST network. Thus, they are already familiar with this paradigm and can easily adapt it to the program of RT sessions proposed here. This project's field collaborator in the Missoula area, The Goodman Group, is eager to be trained and to set up this RT paradigm in their Missoula and Hamilton, Montana facilities.

Data Collection:

PWMLs, assisted by caregivers as necessary, will complete the measures described below three times: 1) prior to the beginning of RT trials, 2) after the 8th week of RT, 3) at the end of the 16-week therapy period. It is estimated that completing these tests will require a total of 70 minutes of time for the PWML and 15-30 minutes for the caregiver.

Summary of Measures:

1. Measure: Cognitive stimulation/reminiscence. Instrument: Autobiographical Memory Interview (AMI), Kopelman, Wilson, and Baddeley, 1989
2. Measure: Dementia severity Instruments: Saint Louis University Mental Status (SLUMS), Tariq, Tumosa, Chibnall, Perry, 2006 Revised Memory and Behavior Problems Checklist (R-MBPC), Teri, Truax, Logsdon, Uomoto, Zarit, Vitaliano, 1992
3. Measure: Social engagement Instrument: Pleasant Events Schedule-AD (PES-AD), Lodsdon, Teri, 1997
4. Measure: Mood Instrument: Geriatric Depression Scale (GDS), van Marwijk, Wallace, de Bock, 1995
5. Measure: Quality of life Instrument: Dementia Quality of Life (DQoL), Brod, Stewart, Sands, Walton, 1999

Interviews. At the end of the 16-week period, interviews will be conducted with all participating RT therapists and with a sample of 15-20 PWMLs who reported the greatest increase in quality of life during the 16 week therapy period. A stratified sampling approach will be used to select the PWMLs for interviews and will consider dementia severity and racial or ethnic background. The experiences of RT therapists and PWMLs with using the 3D printed objects in RT sessions and the online and mobile tools, will be assessed with both structured and open-ended questioning.

ELIGIBILITY:
Inclusion Criteria:

1. English speaking
2. Physician diagnosis of early-stage Alzheimer's disease or mild cognitive impairment
3. Score of 10 or above on the brief St. Louis University Mental Status examination (SLUMS).

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Cognitive stimulation/reminiscence | Will be administered at Week 0 (prior to first therapy session) to establish a baseline. Measures at Week 8 (midpoint of therapy sessions), and Week 16 (following last therapy session) will determine change from the baseline.
  The Autobiographical Memory Interview (AMI) will be completed with PWMLs, a well-established method for assessing autobiographical memory (Kopelman, Wilson, Baddeley, 1989). Specifically, the AMI assesses the extent to which the PWML can recall memories related to factual, incident-specific information from their past. Higher scores indicate greater memory function. An audio recording will be made of the sessions. Later, a written verbal protocol record of each memory produced in the test session will be made from the audio recordings. These verbal protocol records each will be scored independently by two of our researchers. Scoring will be for richness and detail of the reminiscence and will follow the scoring guidelines provided in Kopelman, Wilson, and Baddeley [10]. Inter-rater reliability will be computed. Note that only one measure or score of reminiscence results from the AMI.

SECONDARY OUTCOMES:
Change in Dementia severity-SLUMS | Will be administered at Week 0 (prior to first therapy session) to establish a baseline. Measures at Week 8 (midpoint of therapy sessions), and Week 16 (following last therapy session) will determine change from the baseline.
  The primary measure of dementia severity will be the Saint Louis University Mental Status (SLUMS) (Tariq, Tumosa, Chibnall, Perry, 2006). The SLUMS has 11 items, the scores on which are summed together to produce a total score. The maximum possible score is 30. Normal range for high school educated persons is 27-30 and for less than high school education is 25-30. Mild Neurocogntive Disorder is indicated by scores from 21-26 for high school educated persons and 20-24 for persons with less than high school education. Dementia is indicated by scores from 1-20 for high school educated persons and 1-19 for persons with less than high school education.
Change in Dementia severity-Frequency of Behavioral Problems | Will be administered at Week 0 (prior to first therapy session) to establish a baseline. Measures at Week 8 (midpoint of therapy sessions), and Week 16 (following last therapy session) will determine change from the baseline.
  The Revised Memory and Behavior Problems Checklist (R-MBPC) (Teri, Truax, Logsdon, Uomoto, Zarit, Vitaliano,1992) is a 24-item, caregiver-report measure of observable behavioral problems in dementia patients. It provides "yes-no" scores ("observed" or "not observed") for occurance of patient problems in 3 areas, memory, depression, and disruptive behaviors. It provides a second score for each item reflecting severity of the observed behavior, using a scale of 0-4. The Memory subscale has 7 items. Scores for each item are summed to give a possible subscale score range of 0-7 on occurance of the behavior and 0-28 on severity. Scores on the 9-item depression subscale are summed in the same way, giving a range from 0-9 on observed occurance and 0-36 on severity. The third subscale, Disruptive Behaviors, has 8 items, and when summed across the 8 items gives range of 0-8 for observed occurance and 0-32 for severity.
Change in Dementia severity-dependence on assistance | Will be administered at Week 0 (prior to first therapy session) to establish a baseline. Measures at Week 8 (midpoint of therapy sessions), and Week 16 (following last therapy session) will determine change from the baseline.
  The Katz Index of Independence in Activities of Daily Living rates 6 areas of daily living: bathing; dressing; toileting; transferring; continence, feeding. For each area, 1 point is assigned if no supervision, direction, or personal assistance is needed to perform the activity. For each area, a 0 is assigned if the activity can be performed only with supervision, direction, or personal assistance. Highest possible score is 6 indicating patient is independent. Lowest score is 0, indication patient is very dependent.
Change in Social engagement | Will be administered at Week 0 (prior to first therapy session) to establish a baseline. Measures at Week 8 (midpoint of therapy sessions), and Week 16 (following last therapy session) will determine change from the baseline.
  Pleasant Events/Social Engagement. RT therapists will complete the short form of the Pleasant Events Schedule-AD (PES-AD) for PWMLs (Logsdon and Teri, 1997). The PES-AD short form includes 20 items of events and activities for PWMLs. Items are rated according to their frequency during the past month on a 0-2-point scale: not at all (0), a few times (1), or often (2). Items are also rated 0 or 2 according to how much the patient now enjoys the activity: not at all (0), somewhat (1), or a great deal (2). To obtain an overall summary score for frequency of enjoyable activities, a cross-product of frequency and enjoyment is calculated for each item. Each item can have a score of 0-4. It receives a score of 0 if the patient either does not enjoy or hasn't done in the past month. It receives a score of 4 if the patient enjoys the activity a great deal and has done often. The sum of these item scores represents the frequency of pleasant activities during the past month.
Change in Mood | Will be administered at Week 0 (prior to first therapy session) to establish a baseline. Measures at Week 8 (midpoint of therapy sessions), and Week 16 (following last therapy session) will determine change from the baseline.
  The 15-item Geriatric Depression Scale (GDS) will be used to assess depressive symptoms and mood in PWMLs (van Marwijk, Wallace, de Bock, 1995). This is a well-validated tool to measure mood that is specifically designed for the aging population. It has demonstrated reliability and validity for persons with cognitive impairment. Each of the 15 items receives a score of 0 or 1, with 1 being an indication of depression. The 15 item scores are summed into a total score. Possible range is 0-15. A score of 0 to 5 is considered normal. A score greater than 5 suggests depression.
Change in Quality of Life (self-esteem, positive affect, negative affect, and sense of aesthetics) | Will be administered at Week 0 (prior to first therapy session) to establish a baseline. Measures at Week 8 (midpoint of therapy sessions), and Week 16 (following last therapy session) will determine change from the baseline.
  The scale has 29 items across 5 subdomains: Positive Affect (6 items), Negative Affect (11 items), Feelings of Belonging (3 items), Self-esteem (4 items), and Sense of Aesthetics (5 items). Each item is scored on a scale from 1-5, with 1 indicating "not at all" or "never" and 5 indicating "a lot" or "very often". A score is computed for each subdomain by averaging the item scores from the domain. So subdomain scores range from 1 to 5. No overall DQoL score is computed.

OTHER OUTCOMES:
Functionality and usability of 3D printing mobile tools and paradigm for RT | Interviews will be conducted at 16 weeks
  Interviews will be conducted with all participating RT therapists and with a sample of 15-20 PWMLs who reported the greatest increase in autobiographical memory during the 16 week therapy period. A stratified sampling approach will be used to select the PWMLs for interviews and will consider dementia severity and racial or ethnic background. The experiences of caregiver/therapists and PWMLs with using the 3D printed objects in RT sessions and the online and mobile tools, will be assessed with both structured and open-ended questioning. Qualitative data, not quantitative measures, will result from the interviews. This is a standard practice in engineering to gather qualitative feedback on the software application that has been used in the field trial.

CONTACTS AND LOCATIONS:
Overall Officials: Olu Olofinboba, MS, Principal Investigator — Moai Technologies LLC; Marla Berg-Weger, PhD, Study Director — St. Louis University; Keith Anderson, PhD, Study Director — The University of Texas at Arlington
Locations (2):
- United States (2):
  - Saint Louis University, St Louis, Missouri
  - University of Texas Arlington, Arlington, Texas

IPD SHARING:
Plan to Share IPD: Yes
A data set will be archived. It will consist of the pre-, mid-, and post-test scores of each participant on each of the behavioral measures described in Protocol 9800, and an indication of the 3D-RT dosage group (zero, half, full) to which each participant was assigned. Individuals will be associated with their data only by a number. All other participant identifiers will be removed. We will archive no information about the specific 3D objects each participant used in the study because the objects are inherently autobiographical and personal. DataVerse will be used as the data archiving and sharing platform. The RT therapist iPAD application for 3D object specification will be copyrighted. It will be made available by download from the Moai Technologies' 3D-RT web portal at no cost to other researchers in the field. The results of the project will be shared in the Journal of Gerontological Social Work.
Supporting Information: Study Protocol
Time Frame: At the conclusion of the project, approximately November, 2022
Access Criteria: other researchers in the area of Reminiscence Therapy

REFERENCES:
- [Background] Garlinghouse A, Rud S, Johnson K, Plocher T, Klassen D, Havey T, Gaugler JE. Creating objects with 3D printers to stimulate reminiscence in memory loss: A mixed-method feasibility study. Inform Health Soc Care. 2018 Dec;43(4):362-378. doi: 10.1080/17538157.2017.1290640. Epub 2017 Aug 8. PMID 28786714
- [Background] Woods B, Spector A, Jones C, Orrell M, Davies S. Reminiscence therapy for dementia. Cochrane Database Syst Rev. 2005 Apr 18;(2):CD001120. doi: 10.1002/14651858.CD001120.pub2. PMID 15846613
- [Background] Subramaniam P, Woods B. The impact of individual reminiscence therapy for people with dementia: systematic review. Expert Rev Neurother. 2012 May;12(5):545-55. doi: 10.1586/ern.12.35. PMID 22550983
- [Background] Kopelman MD, Wilson BA, Baddeley AD. The autobiographical memory interview: a new assessment of autobiographical and personal semantic memory in amnesic patients. J Clin Exp Neuropsychol. 1989 Oct;11(5):724-44. doi: 10.1080/01688638908400928. PMID 2808661
- [Background] Tariq SH, Tumosa N, Chibnall JT, Perry MH 3rd, Morley JE. Comparison of the Saint Louis University mental status examination and the mini-mental state examination for detecting dementia and mild neurocognitive disorder--a pilot study. Am J Geriatr Psychiatry. 2006 Nov;14(11):900-10. doi: 10.1097/01.JGP.0000221510.33817.86. PMID 17068312
- [Background] Teri L, Truax P, Logsdon R, Uomoto J, Zarit S, Vitaliano PP. Assessment of behavioral problems in dementia: the revised memory and behavior problems checklist. Psychol Aging. 1992 Dec;7(4):622-31. doi: 10.1037//0882-7974.7.4.622. PMID 1466831
- [Background] Logsdon RG, Teri L. The Pleasant Events Schedule-AD: psychometric properties and relationship to depression and cognition in Alzheimer's disease patients. Gerontologist. 1997 Feb;37(1):40-5. doi: 10.1093/geront/37.1.40. PMID 9046704
- [Background] van Marwijk HW, Wallace P, de Bock GH, Hermans J, Kaptein AA, Mulder JD. Evaluation of the feasibility, reliability and diagnostic value of shortened versions of the geriatric depression scale. Br J Gen Pract. 1995 Apr;45(393):195-9. PMID 7612321
- [Background] Brod M, Stewart AL, Sands L, Walton P. Conceptualization and measurement of quality of life in dementia: the dementia quality of life instrument (DQoL). Gerontologist. 1999 Feb;39(1):25-35. doi: 10.1093/geront/39.1.25. PMID 10028768
- [Background] Cotelli M, Manenti R, Zanetti O. Reminiscence therapy in dementia: a review. Maturitas. 2012 Jul;72(3):203-5. doi: 10.1016/j.maturitas.2012.04.008. Epub 2012 May 16. PMID 22607813
- [Background] Huang HC, Chen YT, Chen PY, Huey-Lan Hu S, Liu F, Kuo YL, Chiu HY. Reminiscence Therapy Improves Cognitive Functions and Reduces Depressive Symptoms in Elderly People With Dementia: A Meta-Analysis of Randomized Controlled Trials. J Am Med Dir Assoc. 2015 Dec;16(12):1087-94. doi: 10.1016/j.jamda.2015.07.010. Epub 2015 Sep 1. PMID 26341034
- [Background] Yates LA, Orrell M, Spector A, Orgeta V. Service users' involvement in the development of individual Cognitive Stimulation Therapy (iCST) for dementia: a qualitative study. BMC Geriatr. 2015 Feb 6;15:4. doi: 10.1186/s12877-015-0004-5. PMID 25655940